CLINICAL TRIAL: NCT00441064
Title: A Randomized, Open-label, Blinded Endpoint, Multi-center, Cross-over Study to Evaluate the Effect of High and Low Sodium Diets on Reduction in Mean 24-hour Ambulatory Blood Pressure in Systolic Hypertensive Patients Treated With Aliskiren (300 mg)
Brief Title: Effect of High and Low Sodium Diets on Blood Pressure in Hypertensive Patients Treated With Aliskiren
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100AUS02
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
Keywords: High blood pressure, hypertension, aliskiren, low sodium diet
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet Sequence Low/High Sodium (Experimental): Patients on low sodium diet ( <= 100 mmol/day) for the first 4 weeks and high sodium (>= 200 mmol/day) diet for the next 4 weeks. [with Aliskiren 300 mg]
  Interventions: Drug: Aliskiren
- Diet Sequence High/Low Sodium (Experimental): Patients on high sodium (>= 200 mmol/day) diet for the first 4 weeks and on low sodium diet ( <= 100 mmol/day) for the next 4 weeks. [with Aliskiren 300 mg]
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This study will compare the effects of high and low level sodium (salt) diets on blood pressure in patients with hypertension (high blood pressure) who are taking aliskiren 300 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18-60 years old
* Patients with systolic hypertension who met the 24 hour Ambulatory Blood Pressure Monitoring (ABPM) criteria (ABPM mean daytime Systolic Blood Pressure (SBP) >= 135 mmHg and < 160 mmHg)

Exclusion Criteria:

* Overt heart failure (HF) or a history of heart failure within preceding 6 months.
* Unstable angina pectoris.
* Type 1 or Type 2 diabetes mellitus or abnormal hemoglobin A1c(HbA1c)
* Body mass index (BMI) > 30 kg/m2
* Subjects taking more than 2 antihypertensive medications.
* Use of other investigational drugs within 30 days of the time of enrollment
* Use of Tamsulosin hydrochloride and other alpha blockers.
* Use of Antiarrhythmic drugs, including digoxin.
* History of MI or cardiovascular attack (CVA) within the preceding 6 months.
* History of malignancy of any organ system, treated or untreated, within the past 5 years with the exception of localized basal cell carcinoma of the skin
* Pregnant or nursing (lactating) women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (19):
- United States (19):
  - Novartis US, Orangevale, California
  - Novartis US, Brooklyn Center, Minnesota
  - Novartis US, Butte, Montana
  - Novartis US, Missoula, Montana
  - Novartis US, Lincoln, Nebraska
  - Novartis US, Johnson City, New York
  - Novartis US, Asheboro, North Carolina
  - Novartis US, Shelby, North Carolina
  - Novartis US, Cincinnati, Ohio
  - Novartis US, Kettering, Ohio
  - Novartis US, Downington, Pennsylvania
  - Novartis US, Erie, Pennsylvania
  - Novartis US, Pittsburgh, Pennsylvania
  - Novartis US, Dallas, Texas
  - Novartis US, Kingsport, Texas
  - Novartis US, Bountiful, Utah
  - Novartis US, Salt Lake City, Utah
  - Novartis US, Port Orchard, Washington
  - Novartis US, Madison, Wisconsin

REFERENCES:
- [Result] Weir MR, Yadao AM, Purkayastha D, Charney AN. Effects of high- and low-sodium diets on ambulatory blood pressure in patients with hypertension receiving aliskiren. J Cardiovasc Pharmacol Ther. 2010 Dec;15(4):356-63. doi: 10.1177/1074248410377173. Epub 2010 Sep 27. PMID 20876343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 patients were randomly assigned to one of the two diet sequences: 69 in the low/high and 63 in the high/low diet sequence. After 4 wks on the assigned diet, patients were then crossed over to the other diet. Patients who were on a high sodium diet for the first 4 wks started on a low sodium diet for the next 4 wks vice versa.
Pre-assignment Details: Safety Population (SP) -Included all randomized patients who received at least 1 dose of study medication. Intent-to-treat population (ITT) -All randomized patients who received at least 1 dose of study medication and had at least 1 valid post baseline assessment of primary efficacy variable.
Groups:
- Diet Sequence Low/High Sodium: Patients on low sodium diet ( <= 100 mmol/day) for the first 4 weeks who crossed over to the high sodium (>= 200 mmol/day) diet for the next 4 weeks. [with Aliskiren 300 mg]
- Diet Sequence High/Low Sodium: Patients on high sodium (>= 200 mmol/day) diet for the first 4 weeks and crossed over to the low sodium diet ( <= 100 mmol/day) for the next 4 weeks. [with Aliskiren 300 mg]
Period: Overall Study
Arm/Group | Diet Sequence Low/High Sodium | Diet Sequence High/Low Sodium
Started | 69 | 63
Safety Population (SP) | 69 | 63
Intent-to-treat (ITT) Population | 61 | 57
Completed | 59 | 56
Not Completed | 10 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Abnormal laboratory values | 0 | 2
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0
Not completed — Protocol Deviation | 3 | 2
Not completed — Patient withdrew consent | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Sequence Low/High Sodium | Diet Sequence High/Low Sodium | Total
Number analyzed (Participants) | 69 | 63 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 51.0 (7.16) | 52.1 (7.75) | 51.5 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 25 | 59
  Male | 35 | 38 | 73
MSSBP [Mean (Standard Deviation); unit: mm Hg] — Mean Sitting Systolic Blood Pressure (MSSBP)
  mm Hg | 147.6 (9.21) | 146.2 (8.94) | 146.9 (9.07)
MSDBP [Mean (Standard Deviation); unit: mm Hg] — Mean Sitting Diastolic Blood Pressure (MSDBP)
  mm Hg | 92.7 (9.81) | 93.6 (8.33) | 93.1 (9.11)
MASBP [Mean (Standard Deviation); unit: mm Hg] — Mean Ambulatory Systolic Blood Pressure (MASBP)
  mm Hg | 138.7 (8.30) | 139.1 (8.52) | 138.9 (8.38)
MADBP [Mean (Standard Deviation); unit: mm Hg] — Mean Ambulatory Diastolic Blood Pressure (MADBP)
  mm Hg | 86.6 (6.73) | 87.7 (7.28) | 87.1 (6.99)

OUTCOME MEASURES:

1. Primary Outcome: Mean 24 Hour Ambulatory Systolic Blood Pressure (MASBP) in Systolic Hypertensive Patients Treated With Aliskiren (300 mg) for 4 Weeks on a High Sodium Diet Versus 4 Weeks on a Low Sodium Diet
Description: The primary objective of the study was to assess mean 24 hour ambulatory systolic blood pressure (MASBP) in systolic hypertensive patients treated with aliskiren (300 mg) for 4 weeks on a high sodium diet versus 4 weeks on a low sodium diet. [At week 4 patients crossed over from low to high sodium diet and vice versa for 4 weeks. MASBP for patients on high sodium diet versus low sodium diet was also analyzed at week 8 (4 weeks after crossover).]
Time Frame: Week 4 and week 8 (4 weeks after crossover)
Population: Completers Population: Included all patients who completed both diet periods - high and low sodium diets
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Low Sodium Diet: All patients who were on low sodium (<= 100 mmol/day) diet
- High Sodium Diet: All patients who were on high sodium (>= 200 mmol/day) diet
Arm/Group | Low Sodium Diet | High Sodium Diet
Number analyzed (Participants) | 115 | 115
mm Hg
  Period 1 (4 weeks) | 124.8 (9.12) | 134.7 (11.13)
  Period 2 (next 4 weeks after crossover) | 123.6 (11.69) | 132.5 (10.07)

2. Secondary Outcome: Mean 24 Hour Ambulatory Diastolic Blood Pressure (MADBP) in Systolic Hypertensive Patients Treated With Aliskiren (300 mg) for 4 Weeks on a High Sodium Diet Versus 4 Weeks on a Low Sodium Diet
Description: To evaluate the mean 24 hour ambulatory diastolic blood pressure (MADBP) in systolic hypertensive patients treated with aliskiren (300 mg) for 4 weeks on a high sodium diet versus 4 weeks on a low sodium diet. [At week 4 patients crossed over from low to high sodium diet and vice versa for 4 weeks. MADBP for patients on high sodium diet versus low sodium diet was also analyzed at week 8 (4 weeks after crossover).]
Time Frame: Week 4 and week 8 (4 weeks after crossover)
Population: Completers Population: Included all patients who completed both diet periods - high and low sodium diets
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Low Sodium Diet | High Sodium Diet
Number analyzed (Participants) | 115 | 115
mm Hg
  Period 1 (4 weeks) | 78.5 (7.37) | 85.0 (9.06)
  Period 2 (next 4 weeks after crossover) | 78.3 (9.10) | 83.2 (8.10)

3. Secondary Outcome: Percentage of Responders Defined as MASBP <130 mm Hg or a Decrease From Baseline in MASBP of ≥20 mm Hg in Systolic Hypertensive Patients Treated With Aliskiren (300 mg) for 4 Weeks on a High Sodium Diet Versus 4 Weeks on a Low Sodium Diet
Description: To evaluate the percentage of responders defined as MASBP < 130 mm Hg or a decrease in MASBP from baseline of ≥20 mm Hg in systolic hypertensive patients treated with aliskiren (300 mg) for 4 weeks on a high sodium diet versus 4 weeks on a low sodium diet. [At week 4 patients crossed over from low to high sodium diet and vice versa for 4 weeks. Percent response for patients on high sodium diet versus low sodium diet was also analyzed at week 8 (4 weeks after crossover).]
Time Frame: Week 4 and Week 8 (4 weeks after crossover)
Population: Completers Population: Included all patients who completed both diet periods - high and low sodium diets
Measure: Number; unit: Percentage of responders
Arm/Group | Low Sodium Diet | High Sodium Diet
Number analyzed (Participants) | 115 | 115
Percentage of responders
  Period 1 (4 weeks) - Response | 78.0 | 41.1
  Period 1 (4 weeks) - No response | 20.3 | 58.9
  Period 2 (next 4 weeks after crossover) - Response | 75.0 | 44.1
  Period 2 (next 4 wks after crossover) -No Response | 25.0 | 55.9

ADVERSE EVENTS:
Time Frame: AE's in overall Safety Population (SP) after 8 weeks
Description: Numbers in AE table are by overall diet, not diet sequence. AEs included overall Safety Population. Low Sodium Diet: 126=69 starters+57 after crossover (56 Completed + 1 who received medication but did not complete study); High Sodium Diet: 124=63 starters+61 after crossover (59 Completed + 2 who received medication but did not complete study)
Arm/Group | Low Sodium Diet | High Sodium Diet
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/124
Other Adverse Events (participants affected / at risk) | 3/126 | 8/124
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Sodium Diet (N=126) | High Sodium Diet (N=124)
Headache (Nervous system disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.